CLINICAL TRIAL: NCT01219127
Title: The Regeneration Effects of Derma-PACE Shockwave in Chronic Diabetic Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Ching-Jen Wang, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-0438C; CMRPG880221 (Other Grant/Funding Number: Chang Gung Research Fund/CMRPG880221)
Record Dates: First submitted 2010-10-10; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2009-02

CONDITIONS: Skin Ulcer
Keywords: Hyperbaric oxygen therapy
MeSH Terms: conditions — Skin Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Derma-PACE (Experimental): Pre-treatment evaluations include complete history and physical examination, chemistry and coagulation profiles, detailed past surgical and medical treatments. The local findings of the ulcer are quantitatively assessed using the S(AD) SAD classification (6) including photo-documentation for the size, shape and configuration of the ulcer
  Interventions: Other: Derma-PACE

INTERVENTIONS:
Other: Derma-PACE — ESWT group received derma-PACE shockwave treatment 2 x 1 wk for 3 wks for a total of 6 treatment using derma-PACE dervice (Alpharetta, GA). HBO groups received HBOT daily 5 days a week for 8 weeks or a total of 40 treatments.

SUMMARY:
Management of chronic diabetic foot skin ulcers require multidisciplinary approaches including diabetic control, wound care, antibiotic, shoe wear off-loading, and surgery in selected cases. The results are inconsistent and irregular, and most studies reported unsatisfactory results. Many adjunctive therapies are implemented in the care of chronic diabetic foot ulcers including hyperbaric oxygen therapy (HBO), ultrasound, recombinant human platelet-derived growth factor-BB (rPDGF-BB), vacuum assisted wound closure (VAWC) and acellular matrix. HBO is the most commonly utilized at the investigators institution. Mixed results of HBO in chronic diabetic foot ulcers are reported. Several studies reported that the beneficial effects of HBO, but none showed universal success. Therefore, the development of a new effective method of treatment for chronic diabetic ulcers is extremely valuable. Extracorporeal shockwave therapy (ESWT) acts as mechanotransduction that produces the therapeutic benefits through complex biological pathways including neovascularization and tissue regeneration. ESWT also showed bacteriostatic effects in experiments. Some studies reported the effectiveness of ESWT in acute and chronic soft tissue wounds. Others reported effectiveness of ESWT in chronic ulcers with 50% completely healed with 6 sessions of treatment. With this background, it appears that ESWT may be effective in the treatment of chronic diabetic foot ulcers. The purpose of this study is to evaluate the efficacy of ESWT in chronic foot ulcers, and to compared with that treated with HBO, and to study the molecular and blood flow perfusion before and after ESWT.

DETAILED DESCRIPTION:
【Background and Purpose】Management of chronic diabetic and ulcers require multidisciplinary approaches including diabetic control, wound care, antibiotic, shoe wear off loading, and surgery in selected cases. The results are inconsistent and irregular, and most studies reported unsatisfactory results. Many adjunctive therapies are implemented in the care of chronic skin ulcers including hyperbaric oxygen therapy (HBO), ultrasound, recombinant human platelet-derived growth factor-BB (rPDGF-BB), vacuum assisted wound closure (VAWC) and acellular matrix. HBO is the most commonly utilized at our institution. Mixed results of HBO in chronic skin ulcers are reported. Several studies reported the beneficial effects in chronic skin ulcers, but none showed universal success. Therefore, the development of a new effective method of treatment for chronic skin ulcers is extremely valuable. Wang et al demonstrated that extracorporeal shockwave acts as mechanotransduction that produces the therapeutic benefits through complex biological pathways including neovascularization and tissue regeneration. Gerdesmeyer et al showed bacteriostatic effects of shockwave in experiments. Schaden et al reported the effectiveness of extracorporeal shockwave in acute and chronic soft tissue wounds. Saggini et all reported effectiveness of ESWT in chronic skin ulcers with 50% completely healed within 6 sessions of treatment. However, no working mechanism of ESWT was discussed. With this background, it appears that extracorporeal shockwave may be effective in the treatment of chronic diabetic ulcers. We have conducted a pilot study using orthowave 180 (TRT, Woodstock, GA) in the treatment of chronic ulcers. The preliminary results of a pilot study in 26 patients with 31 ulcers showed healed or >50% improved ulcers in 90%, 10% unchanged and none worse. The results of the pilot study was published by the Journal of Surgical Research 2009; 152: 96-103. The poster exhibit of this study won the 1st place award in the category of tumor and metabolism of the 75th AAOS annual meeting in San Francisco, CA in March 2008. This study continues the research using derma-PACE (derma-pulse acoustic cellular expression). Derma-PACE (Sanuwave, Alpharetta, GA) is a new shockwave device designed for the treatment of diabetic ulcers. The purpose of this study is to evaluate the efficacy and safety of Derma-PACE shockwave device in the treatment of chronic diabetic ulcers, and to compare the results with that of hyperbaric oxygen therapy, and to investigate the blood flow perfusion, histopathological examination and immunohistochemical analysis.

【Patient selection】This study is approved by The Institutional Review Board on Human Studies. The procedures are performed in accordance with the standards of the Ethical Committee and the Declaration of Helsinki in 1975. All patients are required to sign an informed consent prior to participation in the study. The inclusion criteria include patients with recurrent chronic diabetic ulcers of the extremities for longer than 3 months duration. The exclusion criteria include patients with cardiac arrhythmia or pacemaker, pregnancy, skeletal immaturity patients with malignancy, patients with joint sepsis, ulcers around the skull, spine and chest wall, and patients with poor compliance. A power analysis revealed that a sample size of 32 in each group would be required to establish the statistical significance with α = 0.05 and power = 0.8. We anticipate a drop-out rate of 10 to 15% for various reasons during the course of treatment. Therefore, we plan to recruit 100 patients in the study. Patients are randomly divided into two groups with 50 patients in the shockwave group, and 50 patients in the HBO group who are treated with HBOT. All patients receive the same protocol of diabetic control, wound care, antibiotics and corrective shoe wear etc. Pre-treatment evaluations include complete history and physical examination, chemistry and coagulation profiles, detailed past surgical and medical treatments. The ankle-brachial index (AKI) and HBA1C are assessed individually.

【Technical descriptions】 【Shockwave application】The derma-PACE device is set at E2 @ 4 Hz with the energy level at 0.11 mJ/mm² energy flux density. The dosage of shockwave is wound size dependent. The treatment area includes the actual wound area extended 1.0 cm periphery in every direction. The number of pulses = treatment area (cm²) x 8, but in any case at least 500 shocks. The treatment is performed twice/week for a total of 6 treatments.

【Hyperbaric Oxygen Therapy】Patients receive hyperbaric oxygen therapy (HBO) in a sealed multi-place chamber at a pressure of 2.5 atmospheres absolute (ATA). The treatment starts with the compression of air pressure from 1 ATA to 2.5 ATA in 15 minutes. Patients breathe with 100% medical grade O2 with mask for 25 minutes and take off the mask for O2 break for 5 minutes, and then, repeat breathing 100% O2 with mask for another 25 minutes and off mask for O2 break for 5 minutes. At the end of treatment, the chamber air pressure is decompressed from 2.5 ATA with O2 mask to 1 ATA in 15 minutes. Each patient receives HBO daily, five days a week for a total of 40 treatments.

【Evaluation parameters:】The evaluation parameters include clinical assessment, local blood flow perfusion, bacteriological examination, histopathological evaluation and immunohistochemical analysis from the biopsy specimens. The ulcers are quantitatively assessed using the S(AD)SAD classification for the size, shape and configuration with photo-documentation before and after treatment. The neuropathic sensory change of the foot is examined with pin-prick test. The circulatory status of the affected limb is evaluated with digital palpation of the dorsalis pulsation and ultrasound Doppler perfusion scan. Local blood flow perfusion scan, bacterial culture and sensitivity, and biopsy from the periphary of the ulcer including normal skin is performed before and after treatment, and the specimens are subjected to histomorphological examination and immunohistochemicial stain. The data before and after treatment within the same group and the data between the two groups will be analyzed statistically.

【Anticipated work schedules and results:】We estimate to enroll 2 to 3 patients per week, and it will take approximately one year to recruit sufficient number of patients. It will require 12 additional months for follow-up. Therefore, we estimate a total of three years to complete this study. We anticipate favorable results of ESWT in chronic diabetic ulcers. We also anticipate superior results with ESWT over HBO therapy. Furthermore, we anticipate the improvement in local blood flow perfusion, antibacterial effect as well as angiogenesis and tissue regeneration effects after ESWT. This novel method of treatment may bring in a new insight in the management of chronic diabetic ulcers. Shockwave has the potential to cure chronic skin ulcers without surgery and directly benefits thousands of patients who suffer from this disastrous disease.

ELIGIBILITY:
Inclusion Criteria:

1.recurrent chronic diabetic and non-diabetic skin ulcers of the extremities for longer than 3 months duration.

Exclusion Criteria:

1.patients with cardiac arrhythmia or pacemaker, pregnancy, skeletal immaturity patients with malignancy, patients with joint sepsis, ulcers around the skull, spine and chest wall, and patients with poor compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
anticipate favorable results of derma-PACE ESWT in chronic diabetic ulcers than HBO | 24 month
  We anticipate a favorable result with derma-PACE ESWT compared to HBO. This novel method of treatment may bring in a new insight in the management of chronic diabetic ulcers. Shockwave has the potential to cure chronic diabetic ulcers without surgery and directly benefits thousands of patients who suffer from this disastrous disease.